CLINICAL TRIAL: NCT02999984
Title: Efficacy and Safety of Cryopreserved Formulation of Autologous CD34+ Hematopoietic Stem Cells Transduced Ex Vivo With Elongation Factor 1 Alpha Shortened (EFS) Lentiviral Vector Encoding for Human ADA Gene in Subjects With Severe Combined Immunodeficiency Due to ADA Deficiency
Brief Title: Efficacy and Safety of the Cryopreserved Formulation of OTL-101 in Subjects With ADA-SCID
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: California Institute for Regenerative Medicine (CIRM) (Other); Orchard Therapeutics (Industry)
Responsible Party: Principal Investigator, Donald B. Kohn, M.D., Principal Investigator, University of California, Los Angeles
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OTL-101-4
Record Dates: First submitted 2016-12-19; First posted 2016-12-21 (Estimated); Results first posted 2022-07-22 (Actual); Last update posted 2022-08-03 (Actual); Status verified 2022-08

CONDITIONS: Severe Combined Immunodeficiency Due to ADA Deficiency
Keywords: gene therapy; hematopoietic and progenitor cells; lentiviral vector; ADA-SCID
MeSH Terms: conditions — Severe combined immunodeficiency due to adenosine deaminase deficiency | interventions — Busulfan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes

ARMS (1):
- Gene Therapy (Experimental): Infusion of autologous cryopreserved EFS-ADA LV CD34+ cells
  Interventions: Genetic: Infusion of autologous cryopreserved EFS-ADA LV CD34+ cells (OTL-101); Drug: busulfan; Drug: PEG-ADA ERT

INTERVENTIONS:
Genetic: Infusion of autologous cryopreserved EFS-ADA LV CD34+ cells (OTL-101) — autologous cryopreserved EFS-ADA LV CD34+ cells (OTL-101) are infused intravenously
  Other Names: OTL-101
Drug: busulfan — Busulfan is used for non-myeloablative conditioning
Drug: PEG-ADA ERT — PEG-ADA ERT is discontinued at Day +30 (-3/+15 days) after successful engraftment

SUMMARY:
This is a prospective, non-randomized, single-cohort, longitudinal, single-center, clinical study designed to assess the efficacy and safety of a cryopreserved formulation of OTL-101 (autologous CD34+ hematopoietic stem/progenitor cells transduced ex vivo with EFS (Elongation Factor 1α Short form) Lentiviral Vector (LV) encoding for the human ADA gene) administered to ADA-SCID subjects between the ages of 30 days and 17 years of age, who are not eligible for an Human Leukocyte Antigen (HLA) matched sibling/family donor and meeting the inclusion/exclusion criteria. The OTL-101 product is infused after a minimal interval of at least 24 hours following the completion of reduced intensity conditioning. For subjects who successfully receive the OTL-101 product, pegademase bovine (PEG-ADA) Enzyme Replacement Therapy (ERT) is discontinued at Day+30 (-3/+15) after the transplant. After their discharge from hospital, the subjects will be seen at regular intervals to review their history, perform examinations and draw blood samples to assess immunity and safety.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of written informed consent prior to any study related procedures. In this study consent must be provided by the parents/legal guardians and, where applicable according to local laws, a signed assent from the child,
2. Subjects ≥30 days and <18 years of age,
3. With a diagnosis of ADA-SCID based on:

   Evidence of ADA deficiency, defined as:

   i. Decreased ADA enzymatic activity in erythrocytes, leukocytes, skin fibroblasts, or in cultured fetal cells to levels consistent with ADA-SCID as determined by the reference laboratory, or ii. Identified mutations in ADA alleles consistent with a severe reduction in ADA activity,

   Evidence of ADA-SCID based on either:

   i. Family history of a first order relative with ADA deficiency and clinical and laboratory evidence of severe immunologic deficiency, or ii. Evidence of severe immunologic deficiency in subjects prior to the institution of immune restorative therapy, based on
   * Lymphopenia (absolute lymphocyte count (ALC) <400 cells/µL) OR absence or low number of T cells (absolute CD3+ count < 300 cells/µL), or
   * Severely decreased T lymphocyte blastogenic responses to phytohemagglutinin (either <10% of lower limit of normal controls for the diagnostic laboratory, or <10% of the response of the normal control of the day, or stimulation index <10), or
   * Identification of SCID by neonatal screening revealing low T cell Receptor Excision Circle (TREC) levels.
4. Ineligible for matched family allogeneic Bone Marrow (BM) transplantation, defined as the absence of a medically eligible HLA-identical sibling or family donor, with normal immune function, who could serve as an allogeneic bone marrow donor.
5. Females of child-bearing age will be required to provide a negative pregnancy test 30 days prior to Visit 2.
6. Subjects and their parents/legal guardians must be willing and able to comply with study restrictions and to remain at the clinic for the required duration during the study period and willing to return to the clinic for the follow up evaluation as specified in the protocol.

Exclusion Criteria:

1. Ineligible for autologous Hematopoietic Stem Cell Transplantation (HSCT) as per clinical site criteria.
2. Other conditions which in the opinion of the Principal Investigator and/or Co Investigators, contraindicate the harvest of bone marrow, the administration of Busulfan and the infusion of transduced cells, or which indicate an inability of the subject or subject's parent/legal guardian to comply with the protocol.
3. Hematologic abnormality, defined as:

   * Anemia (Hb <8.0 g/dl).
   * Neutropenia (ANC <500/mm3). Note: ANC <500 with absence of myelodysplastic syndrome on bone marrow aspirate and biopsy and normal marrow cytogenetics are acceptable for eligibility.
   * Thrombocytopenia (platelet count <50,000/mm3, at any age).
   * Prothrombin time or international normalized ratio (INR) and partial thromboplastin time (PTT) >2 x upper limit of normal (ULN) (subjects with a correctable deficiency controlled on medication will not be excluded).
   * Cytogenetic abnormalities on peripheral blood or bone marrow or amniotic fluid (if available).
   * Prior allogeneic HSCT with cytoreductive conditioning.
4. Pulmonary abnormality, defined as:

   * Resting O2 saturation by pulse oximetry <90% on room air.
   * Chest X-ray indicating active or progressive pulmonary disease. Note: Chest X ray indicating residual signs of treated pneumonitis is acceptable for eligibility.
5. Cardiac abnormality, defined as:

   * Abnormal ECG indicating cardiac pathology.
   * Uncorrected congenital cardiac malformation with clinical symptoms.
   * Active cardiac disease, including clinical evidence of congestive heart failure, cyanosis, hypotension.
   * Poor cardiac function as evidenced by left ventricular ejection fraction <40% on echocardiogram.
6. Neurologic abnormality, defined as:

   * Significant neurologic abnormality revealed by examination.
   * Uncontrolled seizure disorder.
7. Renal abnormality, defined as:

   * Renal insufficiency: serum creatinine ≥1.2 mg/dl (106 µmol/L), or ≥3+ proteinuria.
   * Abnormal serum sodium, potassium, calcium, magnesium or phosphate levels at >2 x ULN.
8. Hepatic/gastrointestinal abnormality, defined as:

   * Serum transaminases >5 x ULN.
   * Serum bilirubin >2 x ULN.
   * Serum glucose >1.5 x ULN.
9. Oncologic disease, defined as:

   * Evidence of active malignant disease other than dermatofibrosarcoma protuberans (DFSP).
   * Evidence of DFSP expected to require anti-neoplastic therapy within the 5 years following the infusion of genetically corrected cells (if anti-neoplastic therapy has been completed, a subject with a history of DFSP can be included).
   * Evidence of DFSP expected to be life limiting within the 5 years following the infusion of genetically corrected cells.
10. Known sensitivity to Busulfan.
11. Confirmation of an infectious disease by deoxyribonucleic acid (DNA) Polymerase chain reaction (PCR) positive at time of screening assessment for the following:

    * HIV-1,
    * Hepatitis B,
    * Parvovirus B19.
12. The subject is pregnant or has a major congenital anomaly.
13. Is likely to require treatment during the study with drugs that are not permitted by the study protocol.
14. The subject has previously received another form of gene therapy.

Ages: 30 Days to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Actual)
Dates: Start 2016-12-16 (Actual); Primary Completion 2018-10-11 (Actual); Study Completion 2019-09-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Donald B. Kohn, MD, Study Director — University of California, Los Angeles
Locations (1):
- University of California, Los Angeles, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Carbonaro DA, Zhang L, Jin X, Montiel-Equihua C, Geiger S, Carmo M, Cooper A, Fairbanks L, Kaufman ML, Sebire NJ, Hollis RP, Blundell MP, Senadheera S, Fu PY, Sahaghian A, Chan RY, Wang X, Cornetta K, Thrasher AJ, Kohn DB, Gaspar HB. Preclinical demonstration of lentiviral vector-mediated correction of immunological and metabolic abnormalities in models of adenosine deaminase deficiency. Mol Ther. 2014 Mar;22(3):607-622. doi: 10.1038/mt.2013.265. Epub 2013 Nov 20. PMID 24256635
- [Background] Kohn DB, Booth C, Shaw KL, Xu-Bayford J, Garabedian E, Trevisan V, Carbonaro-Sarracino DA, Soni K, Terrazas D, Snell K, Ikeda A, Leon-Rico D, Moore TB, Buckland KF, Shah AJ, Gilmour KC, De Oliveira S, Rivat C, Crooks GM, Izotova N, Tse J, Adams S, Shupien S, Ricketts H, Davila A, Uzowuru C, Icreverzi A, Barman P, Campo Fernandez B, Hollis RP, Coronel M, Yu A, Chun KM, Casas CE, Zhang R, Arduini S, Lynn F, Kudari M, Spezzi A, Zahn M, Heimke R, Labik I, Parrott R, Buckley RH, Reeves L, Cornetta K, Sokolic R, Hershfield M, Schmidt M, Candotti F, Malech HL, Thrasher AJ, Gaspar HB. Autologous Ex Vivo Lentiviral Gene Therapy for Adenosine Deaminase Deficiency. N Engl J Med. 2021 May 27;384(21):2002-2013. doi: 10.1056/NEJMoa2027675. Epub 2021 May 11. PMID 33974366
- See also: Pre-clinical activity and safety data — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC3944341/

RESULTS

PARTICIPANT FLOW:
Groups:
- Gene Therapy: Infusion of autologous cryopreserved CD34+ cells genetically modified by the EF1αS-ADA (EFS-ADA) lentiviral vector (LV)
  Busulfan: Busulfan is used for non-myeloablative conditioning
  Polyethylene glycol-modified adenosine deaminase (PEG-ADA): PEG-ADA enzyme replacement therapy (ERT) is discontinued at Day 30 +/- 3 days from date of infusion of OTL-101.
Period: Overall Study
Arm/Group | Gene Therapy
Started | 10
Completed | 9
Not Completed | 1
Not completed — Treatment Failure | 1

BASELINE CHARACTERISTICS:
Arm/Group | Gene Therapy
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 10
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 4
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 6
  Afro-American | 2
  Other | 1
  Unknown | 1
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Treatment Efficacy After Treatment With OTL 101 (6 Months)
Description: Efficacy of OTL-101 treatment at 6 months post OTL-101 infusion based on the following parameters and thresholds:
  1. ADA enzyme activity in erythrocytes above baseline/pretreatment level (i.e., >0 units). ADA enzyme activity is measured to assess the amount of functional gene product produced from the normal ADA transgene delivered by EFS-ADA LV.
  2. Absolute CD3+ T cell counts ≥200 cells/μL. Increase in CD3+ T cell counts is a marker of immune reconstitution.
  3. Granulocyte samples positive for vector sequences by quantitative Polymerase Chain Reaction (PCR) (≥1/10,000 cells). Vector copy number (VCN) in the Peripheral Blood (PB) Granulocytes fraction that was T cell depleted, is a surrogate for amount of engrafted genetically modified Hematopoietic stem cell (HSC) that are producing granulocytes every 3-5 days.
Time Frame: 6 months
Population: The efficacy population was a modified intent-to-treat population and consisted of all evaluable subjects at 6-month post-treatment with OTL-101.
  For outcome measure "% of subjects with CD3+ T-cell count >=200 cells/μL", only 9 subjects were evaluable as data was not available for 1 subject.
Measure: Number; unit: percentage of participants
Arm/Group | Gene Therapy
Number analyzed (Participants) | 10
percentage of participants
  % of subjects with an increase from baseline in RBC ADA activity | 100
  % of subjects with CD3+ T-cell count >=200 cells/μL: number analyzed (Participants) | 9
  % of subjects with CD3+ T-cell count >=200 cells/μL | 100
  % of subjects with detectable gene-marked granulocytes by quantitative PCR >=1/10,000 cells | 90

2. Primary Outcome: Overall Survival (OS) of Subjects Treated With Investigational Medicinal Product (IMP) (1 Year)
Description: Overall survival is defined as the percentage of subjects alive at 12 months post- treatment with cryopreserved OTL-101.
Time Frame: 12 Months
Population: The efficacy population was a modified intent-to-treat population and consisted of all subjects treated with OTL-101 within this study.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Gene Therapy
Number analyzed (Participants) | 9
percentage of participants | 100 [66.37 to 100]

3. Primary Outcome: Event-free Survival (EvFS) of Subjects Treated With Investigational Medicinal Product (IMP) (1 Year)
Description: Event-free survival is defined as the percentage of subjects alive with no "event", an "event" being the resumption of PEG-ADA ERT or the need for a rescue allogeneic Hematopoietic Stem Cell Transplant (HSCT), or death.
Time Frame: 12 Months
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Gene Therapy
Number analyzed (Participants) | 10
percentage of participants
  Percentage event-free at 12 months | 90.00 [55.50 to 99.75]
  Percentage without reinstitution of PEG-ADA by 12 months | 90.00 [55.50 to 99.75]
  Percentage without rescue HSCT by 12 months | 100 [66.37 to 100]

4. Secondary Outcome: OS of Subjects Treated With Investigational Medicinal Product (IMP) (2 Years)
Description: OS is defined as the percentage of subjects alive at 24 months post- treatment with cryopreserved OTL-101.
Time Frame: 24 months
Population: The efficacy population was a modified intent-to-treat population and consisted of all subjects treated with OTL-101 within this study, with the exception of 1 subject who was withdrawn prior to Month 24 timepoint.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Gene Therapy
Number analyzed (Participants) | 9
percentage of participants | 100 [66.37 to 100]

5. Secondary Outcome: EvFS of Subjects Treated With Investigational Medicinal Product (IMP) (2 Years)
Description: Event-free survival is defined as the percentage of subjects alive with no "event", an "event" being the resumption of PEG-ADA ERT or the need for a rescue allogenic Hematopoietic Stem Cell Transplant (HSCT), or death.
Time Frame: 24 months
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Gene Therapy
Number analyzed (Participants) | 10
percentage of participants
  Percentage event-free at 24 months | 90.00 [55.50 to 99.75]
  Percentage without reinstitution of PEG-ADA by 24 months | 90.00 [55.50 to 99.75]
  Percentage without rescue HSCT by 24 months | 100 [66.37 to 100]

6. Secondary Outcome: Change From Baseline in CD3+ T Cell Counts (2 Years)
Description: Immune reconstitution was assessed by change in CD3+ T Cell counts over time.
Time Frame: 24 months
Population: The efficacy population was a modified intent-to-treat population and consisted of all subjects treated with OTL-101 within this study, with the exception of 1 subject who was withdrawn prior to Month 24 timepoint and an additional 1 subject for whom CD3+ T cell count data was not available at the Month 24 timepoint.
Measure: Median (Full Range); unit: cells/μL
Arm/Group | Gene Therapy
Number analyzed (Participants) | 8
cells/μL | 418.5 [-332 to 1976]

7. Secondary Outcome: Severe Infections Excluding First 3 Months After Treatment
Description: The infections of interest in this study were severe infections or opportunistic infectious episodes, defined as infections requiring hospitalization or prolonging hospitalization and/or documented infections by opportunistic pathogens. Infections that took place in the first 3 months of follow-up post treatment were excluded from calculations to avoid possible bias introduced in the data by the effects of conditioning.
Time Frame: 24 months
Population: as for outcome 2
Measure: Number; unit: Infections per person per year
Arm/Group | Gene Therapy
Number analyzed (Participants) | 10
Infections per person per year | 0.12

8. Secondary Outcome: Change From Baseline in Quality of Life Measures (2 Years)
Description: Assessment of quality of life was measured by the Lansky Performance Status Scale. The maximum score on the Lansky Performance Scale is 100 - the child is fully active and able to carry on normal activity with no special care needed. The minimum score is 10 - the child is completely disabled, not even passive play. The scores at baseline (pre-treatment with OTL-101) and scores at Month 24 post-treatment with OTL-101 were compared to establish if there were any changes in the child's score in this timeframe.
Time Frame: 24 months
Population: Quality of life data was available for 7/10 subjects at the Month 24 timepoint there only 7 subjects were included in the analysis for this outcome measure.
Measure: Median (Full Range); unit: Lansky Performance Score
Arm/Group | Gene Therapy
Number analyzed (Participants) | 7
Lansky Performance Score | 0 [0 to 0]

9. Secondary Outcome: Percentage of Patients Who Stopped Immunoglobulin Replacement Therapy (IgRT) (2 Years)
Description: Use of immunoglobulin replacement therapies prior to and after gene therapy were monitored. Indications for considering the discontinuation of immunoglobulin replacement therapy included: absolute CD4+ >200, absolute B cell >100/μl, IgA or IgM > lower limit of normal for age or gene marking >1% detectable in B cells.
Time Frame: 24 months
Measure: Number; unit: percentage of participants
Arm/Group | Gene Therapy
Number analyzed (Participants) | 9
percentage of participants | 78

10. Secondary Outcome: Time to Cessation of IgRT for Those Who Stopped (2 Years)
Description: Use of immunoglobulin replacement therapies prior to and after gene therapy were monitored. For subjects who stopped IgRT during the study, the time of cessation was recorded.
Time Frame: 24 months
Population: IgRT data was available for 7/10 subjects at the Month 24 timepoint there only 7 subjects were included in the analysis for this outcome measure.
Measure: Median (Full Range); unit: months
Arm/Group | Gene Therapy
Number analyzed (Participants) | 7
months | 11.6 [9 to 20]

ADVERSE EVENTS:
Time Frame: Adverse events were reported from the time of participant consent, approximately 1-month pre-treatment, up until 2-years post-treatment with OTL-101.
Description: The safety population consisted of all subjects treated with OTL-101 within this study.
Arm/Group | Gene Therapy
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 3/10
Other Adverse Events (participants affected / at risk) | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gene Therapy (N=10)
Bacteraemia (Infections and infestations) | 1 (1)
Bronchiolitis (Infections and infestations) | 1 (1)
Respiratory tract infection viral (Infections and infestations) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gene Therapy (N=10)
Leukopenia (Blood and lymphatic system disorders) | 10 (19)
Neutropenia (Blood and lymphatic system disorders) | 10 (17)
Anaemia (Blood and lymphatic system disorders) | 8 (10)
Thrombocytopenia (Blood and lymphatic system disorders) | 3 (3)
Monocytopenia (Blood and lymphatic system disorders) | 1 (1)
Viral upper respiratory tract infection (Infections and infestations) | 4 (5)
Upper respiratory tract infection (Infections and infestations) | 3 (5)
Otitis media (Infections and infestations) | 3 (4)
Conjunctivitis (Infections and infestations) | 1 (2)
Gastroenteritis (Infections and infestations) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 1 (1)
H1N1 influenza (Infections and infestations) | 1 (1)
Hordeolum (Infections and infestations) | 1 (1)
Respiratory syncytial virus infection (Infections and infestations) | 1 (1)
Tinea infection (Infections and infestations) | 1 (1)
Viral infection (Infections and infestations) | 1 (1)
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 6 (9)
Eczema (Skin and subcutaneous tissue disorders) | 2 (2)
Skin lesion (Skin and subcutaneous tissue disorders) | 1 (2)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1)
Miliaria (Skin and subcutaneous tissue disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 5 (8)
Alanine aminotransferase increased (Investigations) | 5 (6)
Human rhinovirus test positive (Investigations) | 2 (2)
Blood pressure increased (Investigations) | 1 (1)
Haematocrit decreased (Investigations) | 1 (1)
Mean cell haemoglobin concentration decreased (Investigations) | 1 (1)
Mean cell haemoglobin decreased (Investigations) | 1 (1)
Mean cell volume decreased (Investigations) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 5 (8)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 3 (6)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 2 (3)
Vomiting (Gastrointestinal disorders) | 2 (3)
Constipation (Gastrointestinal disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 1 (1)
Retching (Gastrointestinal disorders) | 1 (1)
Pyrexia (General disorders) | 2 (2)
Gait disturbance (General disorders) | 1 (1)
Eye discharge (Eye disorders) | 1 (1)
Eye pruritus (Eye disorders) | 1 (1)
Lacrimation increased (Eye disorders) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Skin abrasion (Injury, poisoning and procedural complications) | 1 (1)
Cerumen impaction (Ear and labyrinth disorders) | 1 (1)
Sinus operation (Surgical and medical procedures) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-03-28): https://cdn.clinicaltrials.gov/large-docs/84/NCT02999984/Prot_000.pdf
  • Statistical Analysis Plan (2018-01-25): https://cdn.clinicaltrials.gov/large-docs/84/NCT02999984/SAP_001.pdf